CLINICAL TRIAL: NCT03319316
Title: Randomized Phase II Study of Durvalumab and Tremelimumab Combination Versus Standard of Care Following First-line Platinum Based Chemotherapy in Two Cohorts of Patients With Non Squamous and Squamous Non-small-cell Lung Cancer (NSCLC)
Brief Title: Combination of Durvalumab and Tremelimumab as Maintenance Treatment in Patients With Non Squamous and Squamous (NSCLC)
Acronym: SOLUTION
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Interest withdrawn
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EORTC-1643; 2017-001827-39 (EudraCT Number)
Record Dates: First submitted 2017-10-16; First posted 2017-10-24 (Actual); Last update posted 2022-01-10 (Actual); Status verified 2021-12

CONDITIONS: Squamous Non-small Cell Lung Cancer; Non-Squamous Non-small Cell Lung Cancer
MeSH Terms: interventions — durvalumab; tremelimumab

STUDY DESIGN:
Intervention Model Description: 2-arm open-label randomized study in each of two separate cohorts (non-squamous and squamous NSCLC) according to histology.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Cohort 1 - Non-squamous - Arm A (Experimental): Patients receive a maintenance treatment of durvalumab + tremelimumab
  Interventions: Drug: Durvalumab; Drug: Tremelimumab
- Cohort 1 - Non-squamous - Arm B (No Intervention): Patients receive a maintenance treatment of pemetrexed
- Cohort 2 - Squamous - Arm A (Experimental): Patients receive a maintenance treatment of durvalumab + tremelimumab
  Interventions: Drug: Durvalumab; Drug: Tremelimumab
- Cohort 2 - Squamous - Arm B (No Intervention): Patients will have observation

INTERVENTIONS:
Drug: Durvalumab — Combination of durvalumab + tremelimumab treatment
  Arms: Cohort 1 - Non-squamous - Arm A; Cohort 2 - Squamous - Arm A
Drug: Tremelimumab — Combination of durvalumab + tremelimumab treatment
  Arms: Cohort 1 - Non-squamous - Arm A; Cohort 2 - Squamous - Arm A

SUMMARY:
This is a multicenter, 2-arm open-label, randomized comparative phase II study in each of two separate cohorts (non-squamous NSCLC and squamous NSCLC) according to histology.

DETAILED DESCRIPTION:
Patients will receive four cycles of standard platinum-based doublet chemotherapy. Upon confirmation of response or tumor stabilization, patients will be registered and allocated into two cohorts based on the tumor histology and each cohort will be randomized into two arms. The experimental arm will receive combination of durvalumab + tremelimumab, the other arm is according to standard of care.

The objective of this trial is to evaluate whether a maintenance approach with the combination immunotherapy with durvalumab + tremelimumab improves progression-free survival (PFS) compared to standard of care in patients with advanced NSCLC. Each cohort is powered separately based on PFS.

ELIGIBILITY:
Inclusion Criteria:

* For inclusion in the study, patients should fulfill the following criteria

  * Histological diagnosis of NSCLC; for non-squamous NSCLC: no known sensitizing EGFR-mutation, no known EML4-ALK translocation. When a patient with non-squamous NSCLC has a KRAS mutation, further testing for EGFR and EML4-ALK is not necessary. For squamous NSCLC, EGFR and EML4-ALK testing is not necessary.
  * Availability of adequate in quality and quantity archived tumor material for IHC PD-L1 testing; (Preferably 15 but 8 mandatory slides or block of tumor tissue will be collected);
  * Stage IIIB or IIIC not eligible for radical treatment or stage IV according to TNM8 (Ref. 6);
  * Brain metastases should be treated with local therapy (stereotactic radiotherapy or whole brain radiotherapy), and patients should be asymptomatic, without treatment with steroids for four weeks before enrollment. Before enrollment, new brain imaging (contrast-CT or gadolinium-MRI) is needed to demonstrate that there is no progression in the brain when the last brain imaging is more than four weeks earlier. Screening for brain metastases is not necessary in patients that were previously not diagnosed with brain metastases and that are without signs indicative of brain metastases.
  * ≥ 18 years of age at time of study entry;
  * WHO performance status 0 or 1; at enrollment
  * Body weight > 30 kg at enrollment
  * Evaluable disease with CT or MRI according to RECIST 1.1 (except for patients with a CR after 4 cycles of platinum-based doublet chemotherapy, these patients are also eligible);
  * Stable disease or response by RECIST criteria response after 4 cycles of platinum-based doublet chemotherapy;
  * Adequate normal organ and marrow function:
  * Absolute neutrophil count (ANC) ≥ 1.5 x 109/L (> 1500 per mm3)
  * Platelet count ≥ 100 x 109/L (>100,000 per mm3)
  * Serum bilirubin ≤ 1.5 x institutional upper limit of normal (ULN). This will not apply to subjects with confirmed Gilbert's syndrome (persistent or recurrent hyperbilirubinemia that is predominantly unconjugated in the absence of hemolysis or hepatic pathology)AST (SGOT)/ALT (SGPT) ≤ 2.5 x institutional upper limit of normal; for patients with liver metastases ≤ 5 x institutional upper limit of normal
  * Measured or calculated creatinine clearance ≥45 mL/min by the Cockcroft-Gault formula (Appendix E)
  * Haemoglobin ≥ 9.0 g/dL
  * Patient with following autoimmune or inflammatory disorders are eligible:
  * Vitiligo or alopecia
  * Hypothyroidism (eg, following Hashimoto syndrome) stable on hormone replacement
  * Any chronic skin condition that does not require systemic therapy
  * Active disease in the last 5 years may be included but only after consultation with the study investigator
  * Celiac disease controlled by diet alone
  * Patient with history of another primary malignancy are eligible in the following cases:
  * Malignancy treated with curative intent and with no known active disease ≥5 years before the first dose of IP and of low potential risk for recurrence
  * Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease
  * Adequately treated carcinoma in situ without evidence of disease
  * Women of child bearing potential (WOCBP) must have a negative serum pregnancy test within 72 hours prior to the first dose of study treatment.

Note: women of childbearing potential are defined as premenopausal females capable of becoming pregnant (i.e. females who have had any evidence of menses in the past 12 months, with the exception of those who had prior hysterectomy). However, women who have been amenorrheic for 12 or more months are still considered to be of childbearing potential if the amenorrhea is possibly due to prior chemotherapy, antiestrogens, low body weight, ovarian suppression or other reasons.

* Patients of childbearing / reproductive potential should use adequate birth control measures, as defined by the investigator, during the study treatment period and from screening to 90 days after the last dose of durvalumab monotherapy or 180 days after the last dose of durvalumab + tremelimumab combination. A highly effective method of birth control is defined as a method which results in a low failure rate (i.e. less than 1% per year) when used consistently and correctly. Such methods include:
* Combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation (oral, intravaginal, transdermal)
* Progestogen-only hormonal contraception associated with inhibition of ovulation (oral, injectable, implantable)
* Intrauterine device (IUD)
* Intrauterine hormone-releasing system (IUS)
* Bilateral tubal occlusion
* Vasectomized partner
* Sexual abstinence (the reliability of sexual abstinence needs to be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the patient)
* Female subjects who are breast feeding should discontinue nursing prior to the first dose of study treatment, from screening to 90 days after the last dose of durvalumab monotherapy or 180 days after the last dose of durvalumab + tremelimumab combination therapy or pemetrexed.
* Subject is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up;
* Before patient registration, written informed consent must be given according to ICH/GCP, and national/local regulations.

Exclusion Criteria:

* Patients should not enter the study if any of the following exclusion criteria is fulfilled

  * Concurrent enrollment in another clinical study, unless it is an observational (non-interventional) clinical study or the follow-up period of an interventional study
  * Mixed small-cell lung cancer and NSCLC histology, sarcomatoid variant or large cell neuro-endocrine variant
  * Patients with known history of leptomeningeal carcinomatosis
  * Any unresolved toxicity NCI CTCAE Grade ≥2 from previous anticancer therapy with the exception of alopecia, vitiligo, and the laboratory values defined in the inclusion criteria
  * Patients with Grade ≥2 neuropathy will be evaluated on a case-by-case basis after consultation with the study investigator
  * Patients with irreversible toxicity not reasonably expected to be exacerbated by treatment with durvalumab or tremelimumab may be included only after consultation with the study investigator
  * Any previous treatment with a PD1 or PD-L1 inhibitor, including durvalumab, a CTLA-4 including tremelimumab or other checkpoint inhibitors or other immune therapy during the last 12 months
  * Current or prior use of immunosuppressive medication within 14 days before the first dose of durvalumab and tremelimumab, with the exceptions of intranasal and inhaled corticosteroids or systemic corticosteroids at physiological doses, which are not to exceed 10 mg/day of prednisone, or an equivalent corticosteroid, or steroids as premedication for hypersensitivity reactions (eg, CT scan premedication)
  * Radiotherapy treatment to more than 30% of the bone marrow or with a wide field of radiation within 4 weeks of the first dose of study drug. Note: Local treatment of isolated lesions, excluding target lesions, for palliative intent is acceptable when it is not within 7 days of the first dose of study drug.
  * Major surgical procedure (as defined by the study investigator) within 28 days prior to the first dose of IP. Note: Local surgery of isolated lesions for palliative intent is acceptable
  * History of allogenic organ transplantation
  * Receipt of live attenuated vaccination within 30 days prior to enrollement
  * Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease [eg, colitis or Crohn's disease], diverticulitis [with the exception of diverticulosis], systemic lupus erythematosus, Sarcoidosis syndrome, or Wegener syndrome [granulomatosis with polyangitis, Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, etc]).
  * History of hypersensitivity to durvalumab, tremelimumab or any excipient
  * Uncontrolled intercurrent illness including, but not limited to:
  * Active infection including tuberculosis (clinical evaluation that includes clinical history, physical examination and radiographic findings, and TB testing in line with local practice), hepatitis B (known positive HBV surface antigen (HBsAg) result), hepatitis C, or human immunodeficiency virus (positive HIV 1/2 antibodies). Patients with a past or resolved HBV infection (defined as the presence of hepatitis B core antibody [anti-HBc] and absence of HBsAg) are eligible. Patients positive for hepatitis C (HCV) antibody are eligible only if polymerase chain reaction is negative for HCV RNA.
  * Symptomatic congestive heart failure, uncontrolled hypertension (defined as blood pressure above 160/90 mm Hg despite medication), unstable angina pectoris, cardiac arrhythmia
  * Active peptic ulcer disease or gastritis
  * Liver cirrhosis CHILD B+, C (Appendix J)
  * Active bleeding diatheses
  * History of primary immunodeficiency
  * Mean QT interval corrected for heart rate (QTc) ≥470 ms calculated from 3 electrocardiograms (ECGs) using Frediricia's Correction
  * Female patients who are pregnant or male or female patients of reproductive potential who are not willing to employ effective birth control from screening to 90 days after the last dose of durvalumab monotherapy or 180 days after the last dose of durvalumab + tremelimumab combination therapy or pemetrexed.
  * Any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule; those conditions should be discussed with the patient before registration in the trial
  * History of another primary malignancy
  * For non-squamous: unable to interrupt aspirin or other nonsteroidal anti-inflammatory agents, other than an aspirin dose <1.3 grams per day, for a 5-day period (8-day period for long-acting agents, such as piroxicam). Unable or unwilling to take folic acid, vitamin B12 supplementation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-11-01 (Estimated); Primary Completion 2021-11 (Estimated); Study Completion 2022-11 (Estimated)

PRIMARY OUTCOMES:
Progression free survival (PFS) | 4.3 years from FPI
  The time interval between the date of randomization and the date of disease progression or death, whichever comes first.

SECONDARY OUTCOMES:
Overall Survival (OS) | 5 years from FPI
  Overall Survival (OS) is defined as the time interval between the date of randomization and the date of death from any cause.
Objective response rate according to RECIST 1.1; | 5 years from FPI
  Patients with response categories progression, early death and unknown will be considered as failing to respond to treatment. The response rates in each arm and their 95% confidence intervals will be provided.
Progression-free survival -2 | 5 years from FPI
  PFS-2 calculated as the time between randomization and the 2nd PD or death, not of the maintenance treatment/observation but the PD after the subsequent treatment thus taking into account the influence of the treatment under investigation on the following treatment line.
Time to failure of 2nd treatment | 5 years from FPI
  Defined as the time between randomization and the permanent treatment interruption of the subsequent/second treatment (treatment received after progression of the first treatment) due to progressive disease, PS worsening, unacceptable toxicity that does not allow continuing the treatment according to the investigator.
Safety | 5 years from FPI
  All adverse events will be recorded according to CTCAE version 4.
Quality of life | 5 years from FPI
  The hypothesis to test is whether the possible benefit with respect to PFS/OS of the intense maintenance treatment will also translate in a better QoL or will the higher risk of Adverse events cause a reduction in QoL. (methodology: quality of life questionnaires)

CONTACTS AND LOCATIONS:
Overall Officials: Martin Reck, Pr, Study Chair — Lungen Clinic Grosshansdorf, Grosshansdorf, Germany; Lizza Hendriks, MD, Study Chair — Academisch Ziekenhuis Maastricht, The Netherlands

IPD SHARING:
Plan to Share IPD: No